CLINICAL TRIAL: NCT04804319
Title: Towards Personalized Dietary Recommendations Based on the Interaction Between Diet, Microbiome and Abiotic Conditions in the Gut
Brief Title: Interactions Between Diet, Microbiome and Abiotic Conditions in the Gut
Acronym: PRIMA
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); KU Leuven (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Henrik Munch Roager, Associate Professor, University of Copenhagen
Other Study IDs: M237
Record Dates: First submitted 2021-03-04; First posted 2021-03-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Diet, Healthy; Metabolic Disease
Keywords: Microbiome; Metabolomics; Nutrition
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 9-days habitual diet — 9-days study with habitual diet including one standardized breakfast on a single day

SUMMARY:
The aim of this study is to explore the interplay between environmental (abiotic) factors in the gut and the gut microbiota composition, diversity and metabolism. Such insights could help us understand personal responses to diets and be a first step towards personalized dietary recommendations targeting the gut microbiome.

DETAILED DESCRIPTION:
The study is a 9-day trial including 85 healthy adults in age between 18 and 75. The participants will throughout the trial register their dietary intake, gastrointestinal symptoms including stool frequency and Bristol stool scale, physical activity, and medicine and supplements intake. Participants will on day 3 and day 5, respectively, consume sweet corns to estimate intestinal transit time by the time it takes sweet corn to travel through the gastrointestinal system. Furthermore, the participants will collect daily urine and stool samples.

On day 2 and day 9, participants will arrive fasting at the department in the morning and have their anthropometry, breath hydrogen and methane levels measured, and a blood sample will be collected from each participant.

The first visit (day 2) also includes a standardized meal test (rye bread, butter, jam, egg, and yogurt with nuts and berries) and intake of paracetamol (250 mg). Subsequently, the participants will stay at the department for the following 6 hours and have their postprandial breath hydrogen and methane measured and urine collected at specific intervals.

Moreover, a sub-set of the participants will on the first visit (day 2) immediately after intake of the standardized meal swallow a single-use gastrointestinal SmartPill capsule, which will monitor their gastrointestinal pH, transit time, temperature and pressure.

ELIGIBILITY:
Inclusion Criteria:

* 18.5-30.0 kg/m2 BMI
* Willing to daily collect a urine and stool sample at home and able to store them in their own freezer in a provided containers throughout the 9-days trial
* Willing to eat sweet corn and report corn-intestinal transit time questionnaire
* Willing to record 9 days dietary intake and defecation pattern
* Willing to have blood samples drawn two times
* Owns a device with access to the internet and is willing to use myfood24 platform
* Known ability to tolerate paracetamol and willing to consume ½ paracetamol tablet dissolved in water (250mg)
* Willing to eat rye bread, butter, jam, egg, yoghurt, berries and nuts

Exclusion Criteria:

* Any condition that makes the project responsible researcher to doubt the feasibility of the volunteer´s participation
* Pregnant or lactating women
* Suffering from inflammatory bowel syndrome (IBS), small intestinal bacterial overgrowth (SIBO) or inflammatory bowel diseases (IBD)
* Intake of antibiotics, diarrhea inhibitors and laxatives ˂ 1month
* Current chronic or infectious diseases
* Diagnosis of diabetes
* History of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
* Frequent intake of painkillers or other medication (mild antidepressants and contraceptive pills are allowed)
* Concurrent participation in another trial

Additional exclusion criteria for the SmartPill sub-study:

* Intake of medications potentially altering gastric pH (proton pump inhibitors, histamine receptor antagonists, antacids)
* Intake of medications potentially altering the gastrointestinal motility (prokinetics, antiemetic agents, anticholinergic agents, narcotic analgetics, nonsteroidal anti-inflammatory drugs)
* Dysphagia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Faecal pH vs gut microbial saccharolytic/proteolytic metabolism | Day 1-9
  We test whether faecal pH is positively associated with microbial-derived proteolytic metabolites (i.e. p-cresol sulfate and phenylacetylglutamine) in urine and negatively associated with microbial-derived saccharolytic metabolites in faeces (i.e. acetate, butyrate and propionate)

SECONDARY OUTCOMES:
Abiotic factors vs faecal metagenomic profile | Day 1-9
  We test whether day-to-day variations in abiotic factors (faecal and/or intestinal pH, faecal redox potential, intestinal transit time and substrate availability) are associated with changes in the faecal microbiome
Abiotic factors vs faecal metabolome | Day 1-9
  We test whether day-to-day variations in abiotic factors (faecal and/or intestinal pH, faecal redox potential, intestinal transit time and substrate availability) are associated with changes in the faecal metabolome
Abiotic factors vs urine metabolome | Day 1-9
  We test whether day-to-day variations in abiotic factors (faecal and/or intestinal pH, faecal redox potential, intestinal transit time and substrate availability) are associated with changes in the urine metabolome
Abiotic factors vs blood metabolome | Day 2 and 9
  We test whether day-to-day variations in abiotic factors (faecal and/or intestinal pH, faecal redox potential, intestinal transit time and substrate availability) are associated with changes in the blood (serum) metabolome
Abiotic factors vs microbial-derived metabolites | Day 1-9
  We test whether day-to-day variations in abiotic factors (faecal and/or intestinal pH, faecal redox potential, intestinal transit time and substrate availability) are associated with changes in diet-derived microbial metabolites in blood/urine/faeces, including short-chain fatty acids, secondary bile acids, phenolic and indolic compounds, branched-chain fatty acids, trimethylamine N-oxide, hippuric acid, urolithin, and enterolactone
Faecal metagenomics profile vs metabolome | Day 1-9
  We test whether day-to-day variations in the microbiome are associated with changes in diet-derived microbial metabolites in blood/urine/faeces, including short-chain fatty acids, secondary bile acids, phenolic and indolic compounds, branched-chain fatty acids, trimethylamine N-oxide, hippuric acid, urolithin, and enterolactone

OTHER OUTCOMES:
Faecal microbiome | Day 1-9
  Determination of the variation in the intra- and inter-individual microbiomes in all faecal samples collected from day 1 to day 9
Faecal metabolome | Day 1-9
  Changes in the faecal metabolome within and between volunteers as determined by untargeted metabolic profiling by liquid chromatography mass spectrometry (LC-MS) of all faecal samples collected from day 1 to day 9
In vitro metabolic profiling | Day 1-9
  Metabolic profiling of in vitro microbial communities inoculated by faecal outputs from the study
Urine metabolome | Day 1-9
  Changes in the urine metabolome within and between volunteers as determined by untargeted metabolic profiling by LC-MS of all urine samples collected from day 1 to day 9
Postprandial urine metabolome | Day 2
  Diet- and microbial-derived metabolites from the standardised meal determined by metabolic profiling by LC-MS of postprandial urine samples collected at 30 min, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 6-8 hours, 8-10 hours, 10-24 hours
Food intake markers | Day 2-3 and day 8-9
  Food intake biomarkers determined by metabolic profiling by LC-MS of 24-hour urine collection at day 2-3 and day 8-9.
Blood metabolome | Day 2 and 9
  Changes in the blood metabolome within and between volunteers as determined by untargeted metabolic profiling by LC-MS of fasting blood samples collected at day 2 and day 9
Fasting breath hydrogen and methane | Day 2 and 9
  Measurement of fasting breath hydrogen and methane exhalation at day 2 and day 9
Postprandial breath hydrogen and methane | Day 2
  Measurement of fasting and postprandial breath hydrogen and methane exhalation after standardized breakfast (every 30 min until 6 hours post-meal)
Plasma levels of short chain fatty acids | Day 2 and day 9
  Measurement of fasting plasma short-chain fatty acids determined by LC-MS from day 2 and day 9
Faecal levels of short chain fatty acids | Day 1-9
  Measurements of short-chain fatty acids in all faecal samples collected from day 1 to day 9 determined by LC-MS
Intestinal transit time | Day 2-7
  1. Whole transit time variation within and between volunteers as determined by the "sweet-corn test". Briefly, participants are instructed to consume sweet corns twice, on day 3 and 5, and to record the times until visible corn excretion on these two occasions, as well as their defecation frequency, and stool consistency during days 1 to 9
  2. Whole transit time variation within and between volunteers as determined by the SmartPill Wireless Motility Capsule in the subgroup
  3. Comparison of the whole intestinal transit time data obtained by the Smartpill Wireless Motility Capsule and results from the sweet-corn test in the subgroup
  4. Small bowel transit time determined by the SmartPill Wireless Motility Capsule in the subgroup
  5. Colonic transit time determined by the SmartPill Wireless Motility Capsule in the subgroup
Gastric emptying | Day 2
  1. Fluid gastric emptying time determined by the presence of paracetamol metabolites in postprandial urine samples
  2. Solid gastric emptying time determined by the SmartPill Wireless Motility Capsule in the subgroup
Appetite hormones | Day 2 and 9
  Determination of different appetite hormones in fasting blood samples at day 2 and day 9 to record baseline values
Glucose levels | Day 2 and 9
  Measurements of glucose in fasting blood samples at day 2 and day 9
Insulin levels | Day 2 and day 9
  Measurement of insulin levels in fasting blood samples at day 2 and day 9
C-peptide levels | Day 2 and day 9
  Measurement of C-peptide levels in fasting blood samples at day 2 and day 9
HbA1c levels | Day 2 and day 9
  Measurement of HbA1c levels in fasting blood samples at day 2 and day 9
Immune system markers | Day 2 and 9
  Measurements of fasting plasma cytokines, C-reactive protein (CRP), lipopolysaccharides (LPS), lipopolysaccharide binding protein (LPS-BP) at day 2 and day 9 to record baseline values
Lipid metabolism | Day 1-9
  Determination of bile acids in fasting blood samples at day 2 and day 9 and in all faecal samples from day 1 to day 9 to associate with changes in abiotic factors
9-days dietary intake | Day 1-9
  Assessment of dietary intake via myfood24 dietary recalls from day 1 to day 9
Faecal nitrogen | Day 1-9
  Assessment of nitrogen in all faecal samples from day 1 to day 9
Faecal residual carbohydrates | Day 1-9
  Assessment of residual carbohydrates in all faecal samples from day 1 to day 9
Faecal energy | Day 1-9
  Assessment of total energy in all faecal samples from day 1 to day 9
Microbial load assessed by qPCR | Day 1-9
  Assessment of microbial load by quantitative PCR in all faecal samples from day 1 to day 9
Microbial load assessed by flow cytometry | Day 1-9
  Assessment of microbial cell counts by flow cytometry in all faecal samples from day 1 to day 9
Faecal pH | Day 1-9
  Measurements of pH in all faecal samples from day 1 to day 9
Faecal redox potential | Day 1-9
  Measurements of redox potential in all faecal samples from day 1 to day 9
Faecal ionic strength | Day 1-9
  Measurements of ionic strength (Na+ and K+) in all faecal samples from day 1 to day 9
Faecal water content | Day 1-9
  Measurements of water content in all faecal samples from day 1 to day 9
Subjective gastrointestinal symptoms | Day 1-9
  Gastrointestinal symptoms reported on a scale from 0 to 10, where 0 means no symptoms and 10 means the worst possible symptoms. The questionnaire includes these symptoms: overall stomach and intestine symptoms, stomachache, flatulence, bloating, constipation, and diarrhea.
Creatinine | Day 2
  Measurements of urinary levels of creatinine from controlled 6-hour urine collection
Intestinal pH | Day 2-7
  pH measurements throughout the gastrointestinal system determined by the SmartPill Wireless Motility Capsule in the subgroup
Intestinal epithelial cell shedding | Day 1-9
  Measurements of host DNA content in all faecal samples from day 1 to day 9

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

REFERENCES:
- [Result] Prochazkova N, Laursen MF, La Barbera G, Tsekitsidi E, Jorgensen MS, Rasmussen MA, Raes J, Licht TR, Dragsted LO, Roager HM. Gut physiology and environment explain variations in human gut microbiome composition and metabolism. Nat Microbiol. 2024 Dec;9(12):3210-3225. doi: 10.1038/s41564-024-01856-x. Epub 2024 Nov 27. PMID 39604623